CLINICAL TRIAL: NCT05846035
Title: Paraneoplastic Syndrome in Hepatocellular Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hala Maher Abdelhafiz, resident of Tropical department, Sohag University
Other Study IDs: Soh-Med-23-04-12MS
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Triphasic C.T abdomen and pelvis — for cirrhotic patients to ensure hepatocellular carcinoma
  Other Names: alpha feto protein

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most common cancer in the world with rising incidence. Globally, there has been substantial variation in prevalence of risk factors for HCC over years, like control of viral hepatitis in developing countries but growing epidemic of fatty liver disease in developed world. Changing epidemiology of HCC is related to trends in these risk factors, Paraneoplastic syndromes (PNS) are defined as systemic, metabolic, or other distant consequences of malignancy resulting, either directly or indirectly, from production by the neoplasm of substances that gain access to the blood stream, thereby exerting their effects on distant organs or tissues There is four major HCC-associated paraneoplastic syndromes among Cirrhotic patients,i.e.hypercholesterolemia,hypoglycemia,hypercalcemia,and erythrocytosis .

ELIGIBILITY:
Inclusion Criteria:

* - Cirrhotic Patients with HCC.
* HCC will be diagnosed based on Alpha -feto protein (AFP) and dynamic imaging.

Exclusion Criteria:

* - Patient known to have primary parathyroid disease, patients with bone metastasis or excessive use of antacids.
* Patients with secondary polycythemia (as chronic hypoxia) and patients with polycythemia rubra vera.
* Patients with acute infections or GIT bleeding.
* Patients with preexisting dyslipidemia.
* Patients with significant cholestasis.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Cirrhotic Patients with HCC.
  * HCC will be diagnosed based on Alpha -feto protein (AFP) and dynamic imaging.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
the prevalence of Paraneoplastic Syndrome in cirrhotic Patients with HCC. | 12 months
  To investigate the prevalence of PNS (hypoglycemia, hypercholesterolemia, hypercalcemia, erythrocytosis, and thrombocytosis) and clinical characteristics in cirrhotic Patients with HCC.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Borde T, Nezami N, Laage Gaupp F, Savic LJ, Taddei T, Jaffe A, Strazzabosco M, Lin M, Duran R, Georgiades C, Hong K, Chapiro J. Optimization of the BCLC Staging System for Locoregional Therapy for Hepatocellular Carcinoma by Using Quantitative Tumor Burden Imaging Biomarkers at MRI. Radiology. 2022 Jul;304(1):228-237. doi: 10.1148/radiol.212426. Epub 2022 Apr 12. PMID 35412368
- [Background] Qu Q, Wang S, Chen S, Zhou L, Rui JA. Prognostic role and significance of paraneoplastic syndromes in hepatocellular carcinoma. Am Surg. 2014 Feb;80(2):191-6. PMID 24480222
- [Background] Samant H, Amiri HS, Zibari GB. Addressing the worldwide hepatocellular carcinoma: epidemiology, prevention and management. J Gastrointest Oncol. 2021 Jul;12(Suppl 2):S361-S373. doi: 10.21037/jgo.2020.02.08. PMID 34422400